CLINICAL TRIAL: NCT00561353
Title: A Blinded, Randomized, Placebo-controlled Trial in Genotype 1 Hepatitis C-Infected Subjects to Evaluate the Efficacy, Safety, Tolerability and Pharmacokinetics of Repeated Doses of TMC435350, With or Without Peginterferon Alpha-2a and Ribavirin
Brief Title: A Study of TMC435350 Administered With or Without Standard of Care Therapy in Participants With Genotype 1 Hepatitis C Virus Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR012607; TMC435350-TiDP16-C201 (Other: Tibotec Pharmaceuticals, Ireland); NCT00614185 (obsolete NCT alias)
Record Dates: First submitted 2007-11-19; First posted 2007-11-20 (Estimated); Results first posted 2014-02-06 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C, Chronic; Tibotec; TMC435350-TiDP16-C201; TMC435350-C201; TMC435; PEGASYS (peginterferon alpha-2a, PegIFNα-2a); COPEGUS (ribavirin)
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Simeprevir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- TMC435 25 mg (Cohort 1/Panel A and B) (Experimental): Treatment-naïve participants received TMC435 25 mg once daily for 7 days followed by TMC435 25 mg once daily coadministered with peginterferon alpha-2a (PegIFNα-2a) (P) and ribavirin (R) for 21 days (Panel A) OR TMC435 25 mg once daily coadministered with PR for 28 days (Panel B).
  Interventions: Drug: TMC435; Drug: Peginterferon (PegIFNα-2a); Drug: Ribavirin
- TMC435 75mg (Cohort 1/Panel A and B) (Experimental): Treatment-naïve participants received TMC435 75 mg once daily for 7 days followed by TMC435 75 mg once daily for 21 days with PegIFNα-2a (P) and ribavirin (R) OR TMC435 75 mg once daily coadministered with PR for 28 days (Panel B).
  Interventions: Drug: TMC435; Drug: Peginterferon (PegIFNα-2a); Drug: Ribavirin
- Placebo (Cohort 1/Panel A and B) (Placebo Comparator): Treatment-naïve participants received placebo (identical in appearance to TMC435 25/75 mg) once daily for 7 days followed by placebo once daily coadministered with PegIFNα-2a (P) and ribavirin (R) for 21 days (Panel A) OR and Placebo once daily coadministered with PR for 28 days (Panel B).
  Interventions: Drug: Placebo; Drug: Peginterferon (PegIFNα-2a); Drug: Ribavirin
- TMC435 200 mg (Cohort 2, Panel A and B) (Experimental): Treatment-naïve participants received TMC435 200 mg once daily for 7 days followed by TMC435 200 mg once daily coadministered with PegIFNα-2a (P) and ribavirin (R) for 21 days (Panel A) OR TMC435 200 mg once daily coadministered with PR for 28 days (Panel B).
  Interventions: Drug: TMC435; Drug: Peginterferon (PegIFNα-2a); Drug: Ribavirin
- Placebo (Cohort 2/Panel A and B) (Placebo Comparator): Treatment-naïve participants received placebo (identical in appearance to TMC435 200 mg) once daily for 7 days followed by placebo once daily coadministered with PegIFNα-2a (P) and ribavirin (R) for 21 days (Panel A) OR placebo once daily coadministered with PR for 28 days (Panel B).
  Interventions: Drug: Placebo; Drug: Peginterferon (PegIFNα-2a); Drug: Ribavirin
- TMC435 75 mg (Cohort 4/Panel C) (Experimental): Treatment-experienced non-responders received TMC435 75 mg once daily coadministered with PegIFNα-2a and ribavirin for 28 days.
  Interventions: Drug: TMC435; Drug: Peginterferon (PegIFNα-2a); Drug: Ribavirin
- TMC435 150 mg (Cohort 4/Panel C) (Experimental): Treatment-experienced non-responders received TMC435 150 mg once daily coadministered with PegIFNα-2a and ribavirin for 28 days.
  Interventions: Drug: TMC435; Drug: Peginterferon (PegIFNα-2a); Drug: Ribavirin
- TMC435 200 mg (Cohort 4/Panel C) (Experimental): Treatment-experienced non-responders received TMC435 200 mg once daily coadministered with PegIFNα-2a and ribavirin for 28 days.
  Interventions: Drug: TMC435; Drug: Peginterferon (PegIFNα-2a); Drug: Ribavirin
- Placebo (Cohort 4/Panel C) (Placebo Comparator): Treatment-experienced non-responders received placebo once daily coadministered with PegIFNα-2a and ribavirin for 28 days.
  Interventions: Drug: Placebo; Drug: Peginterferon (PegIFNα-2a); Drug: Ribavirin
- TMC435 200 mg (Cohort 5/Panel D) (Experimental): Treatment-experienced relapsers received TMC435 200 mg once daily coadministered with PegIFNα-2a and ribavirin for 28 days.
  Interventions: Drug: TMC435; Drug: Peginterferon (PegIFNα-2a); Drug: Ribavirin

INTERVENTIONS:
Drug: TMC435 — TMC435 25 mg, 75 mg, 150 mg, or 200 mg capsules taken orally (by mouth) once daily for 21 or 28 days.
  Arms: TMC435 150 mg (Cohort 4/Panel C); TMC435 200 mg (Cohort 2, Panel A and B); TMC435 200 mg (Cohort 4/Panel C); TMC435 200 mg (Cohort 5/Panel D); TMC435 25 mg (Cohort 1/Panel A and B); TMC435 75 mg (Cohort 4/Panel C); TMC435 75mg (Cohort 1/Panel A and B)
Drug: Placebo — Placebo capsules identical in appearance to TMC435 capsules taken orally (by mouth) once daily for 28 days.
  Arms: Placebo (Cohort 1/Panel A and B); Placebo (Cohort 2/Panel A and B); Placebo (Cohort 4/Panel C)
Drug: Peginterferon (PegIFNα-2a) — One subcutaneous (under the skin) injection containing 0.5 mL solution with 180 mcg PegIFNα-2a on Days 1, 8, 15, and 22
  Other Names: PEGASYS
Drug: Ribavirin — 200-mg tablets of ribavirin (body-weight adjusted dose) taken orally (by mouth) twice daily for 21 or 28 days in Cohorts 1 and 2 and for 28 days in Cohorts 4 and 5.
  Other Names: COPEGUS

SUMMARY:
The purpose of this study is to investigate how efficient TMC435350 will work against the Hepatitis C virus genotype 1 (genotypes refer to the genetic constitution of the virus) and what the concentrations of TMC435350 in the blood are with or without pegylated interferon alpha-2a (PegIFNa-2a) or PegIFNa-2a plus ribavirin.

DETAILED DESCRIPTION:
This is a blinded (participant and study staff will not know the identity of assigned treatments), randomized (participants assigned to treatment by chance), placebo-controlled (a term used to describe a method of research in which an inactive substance referred to as a placebo is given to one group of participants, while the treatment being tested is given to another group) study to assess the effectiveness, safety, tolerability, and pharmacokinetics (to test the concentration of study drug in the blood over time) of different dose regimens of TMC435350 (hereafter referred to as TMC435) given alone or in combination with peginterferon alpha-2a (PegIFNa-2a) and ribavirin. TMC435 is a new drug that is development for the treatment of Hepatitis C virus (HCV) infection and belongs to a class of drugs that work by blocking an enzyme (protease) that the HCV needs to replicate. The combination of PegIFNa-2a and ribavirin are current standard of care (SoC) therapy for patients with chronic HCV infection. Approximately 72 participants with HCV infection who have never been treated for HCV infection (referred to as treatment-naïve participants) and 36 participants who have been treated for HCV infection (referred to as treatment-experienced participants) who did not respond to previous therapy with interferon (IFN) and who did not discontinue previous anti-HCV therapy because of adverse events [AEs]) will be included in this study. Two blinded placebo-controlled groups (referred to as "cohorts") of treatment-naïve participants will be sequentially initiated TMC435 to ensure that a higher dose is only administered if the previous lower dose is found safe and tolerable. The first group (Cohort 1) of treatment-naïve participants will receive low-doses of TMC435 or placebo for 7 days followed by 21 days of combined tritherapy with PegIFNa-2a and ribavirin OR participants will receive 28 days of tritherapy (TMC435 or placebo + PegIFNa-2a and ribavirin). After review of data from Cohort 1, a second group (Cohort 2) of treatment-naïve participants will be given higher doses of TMC435 or placebo in the same manner described for the first cohort. A third group (Cohort 3) of participants previously planned in the study will not be enrolled. After review of data from Cohort 2, a fourth group (Cohort 4) of treatment-experienced participants will be given 28 days of TMC435 (or placebo) as tritherapy with PegIFNa-2a and ribavirin to determine the maximum tolerated dose of TMC435. In addition, up to 10 HCV-infected individuals (who participated in study TMC435350-TiDP16-C101 (ClinicalTrials.gov registry number NCT00938899) will comprise Cohort 5 and will be given 28 days of TMC435 at a dose previously determined to be safe and efficacious as tritherapy with PegIFNa-2a and ribavirin. Blood samples will be taken from participants at protocol-specified time points to determine plasma concentrations of TMC435 and ribavirin and safety will be monitored throughout the study. Individuals will participate in this study for up 54 weeks (includes up to 6 weeks during the screening period followed by up to 4 weeks of study treatment with TMC435 (or placebo) and up to a maximum of 44 weeks of treatment with PegIFNa-2a and ribavirin.

ELIGIBILITY:
Inclusion Criteria: - Documented chronic genotype 1 Hepatitis C infection - Able to comply with the protocol requirements and having good accessible veins - Amount of virus in the blood (HCV RNA) >= 10.000 IU/mL, at screening - Bodyweight as defined by a Quetelet Index (Body Mass Index [BMI]) between 18 and 32 kg/m², extremes included Exclusion Criteria: - Evidence of liver cirrhosis or decompensated liver disease or any other form of non-viral hepatitis - Participants receiving or having received treatment with polymerase inhibitor or protease inhibitor, or Standard of Care therapy with COPEGUS (ribavirin) and PEGASYS (peginterferon alpha-2a) for treatment for HCV during the 6 months before screening - Male participants with female partners of childbearing potential not agreeing to use a reliable birth control method, Female, except if postmenopausal for over 2 years, or posthysterectomy, or post-tubal ligation (without reversal operation) - History or evidence of current use of alcohol, barbiturate, amphetamine, recreational or narcotic drug use, which would compromise the participant 's safety and/or compliance. A positive urine drug test at screening. Urine will be tested to check the current use of amphetamines, cocaine, and opioids (with the exclusion of methadone) - Participants having at least one lab toxicity that is found to be clinically significant - Participants co-infected with HIV, or Hepatitis A or B, or hepatitis B surface antigen, or active tuberculosis at screening, participants with prolonged QTc (>480 ms) value or any cardiac disease at screening, or any active clinically significant disease (e.g., cardiac dysfunction, cardio(myo)pathy, cardiac insufficiency), or medical history or physical examination findings during screening that, in the Investigator's opinion, would compromise the outcome of the trial - Participants having uncontrolled/unstable diabetes, epilepsy, a manifest psychiatric disease, non-stable methadone (or equivalent drug) use or participants having any other unstable disease, participants enrolled in another clinical trial within 90 days prior to screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals, Ireland Clinical Trial, Study Director — Tibotec Pharmaceuticals, Ireland
Locations (24):
- Belgium (4):
  - Bruges
  - Brussels
  - Edegem
  - Ghent
- France (6):
  - Clichy
  - Lyon
  - Marseille
  - Paris
  - Pessac
  - Vandœuvre-lès-Nancy
- Germany (7):
  - Berlin
  - Düsseldorf
  - Freiburg im Breisgau
  - Hamburg
  - Hanover
  - Kiel
  - München
- Amsterdam-Zuidoost, Netherlands
- Poland (4):
  - Bialystok
  - Kielce
  - Lodz
  - Warsaw
- United Kingdom (2):
  - London
  - Plymouth

REFERENCES:
- [Derived] Benguigui L, Le Gouzouguec S, Balanca B, Ristovski M, Putet G, Butin M, Guillois B, Beissel A. A Customizable Digital Cognitive Aid for Neonatal Resuscitation: A Simulation-Based Randomized Controlled Trial. Simul Healthc. 2024 Oct 1;19(5):302-308. doi: 10.1097/SIH.0000000000000790. Epub 2024 Apr 8. PMID 38587329
- [Derived] Lenz O, de Bruijne J, Vijgen L, Verbinnen T, Weegink C, Van Marck H, Vandenbroucke I, Peeters M, Simmen K, Fanning G, Verloes R, Picchio G, Reesink H. Efficacy of re-treatment with TMC435 as combination therapy in hepatitis C virus-infected patients following TMC435 monotherapy. Gastroenterology. 2012 Nov;143(5):1176-1178.e6. doi: 10.1053/j.gastro.2012.07.117. Epub 2012 Aug 8. PMID 22885330
- [Derived] Manns M, Reesink H, Berg T, Dusheiko G, Flisiak R, Marcellin P, Moreno C, Lenz O, Meyvisch P, Peeters M, Sekar V, Simmen K, Verloes R. Rapid viral response of once-daily TMC435 plus pegylated interferon/ribavirin in hepatitis C genotype-1 patients: a randomized trial. Antivir Ther. 2011;16(7):1021-33. doi: 10.3851/IMP1894. PMID 22024518

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 25 sites in 6 countries: Belgium, France, Germany, Poland, the Netherlands, and the United Kingdom.
Pre-assignment Details: A total of 121 participants infected with Hepatitis C virus (HCV) were randomized of whom 116 were treated. Reasons for not receiving treatment were withdrawal of consent (4 participants) and sponsor's decision (1 participant).
Groups:
- TMC435 25 mg (Cohort 1/Panel A and B): Treatment-naïve participants received TMC435 25 mg once daily for 7 days followed by TMC435 25 mg once daily coadministered with ribavirin (RBV) for 21 days + peginterferon alpha-2a (PegIFNα-2a) on Days 8, 15, and 22 (Panel A) OR TMC435 25 mg once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22 (Panel B)
- TMC435 75mg (Cohort 1/Panel A and B): Treatment-naïve participants received TMC435 75 mg once daily for 7 days followed by TMC435 75 mg once daily coadministered with RBV for 21 days + PegIFNα-2a on Days 8, 15, and 22 (Panel A) OR TMC435 75 mg once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22 (Panel B)
- Placebo (Cohort 1/Panel A and B): Treatment-naïve participants received placebo (identical in appearance to TMC435 25 mg or 75 mg) once daily for 7 days followed by placebo once daily coadministered with RBV for 21 days + PegIFNα-2a on Days 8, 15, and 22 (Panel A) OR placebo once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22 (Panel B)
- TMC435 200 mg (Cohort 2, Panel A and B): Treatment-naïve participants received TMC435 200 mg once daily for 7 days followed by TMC435 200 mg once daily coadministered with RBV for 21 days + PegIFNα-2a on Days 8, 15, and 22 (Panel A) OR TMC435 200 mg once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22 (Panel B)
- Placebo (Cohort 2/Panel A and B): Treatment-naïve participants received placebo (identical in appearance to TMC435 200 mg) once daily for 7 days followed by placebo once daily coadministered with RBV for 21 days + PegIFNα-2a on Days 8, 15, and 22 (Panel A) OR placebo once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22 (Panel B)
- TMC435 75 mg (Cohort 4/Panel C): Treatment-experienced non-responders received TMC435 75 mg once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22.
- TMC435 150 mg (Cohort 4/Panel C): Treatment-experienced non-responders received TMC435 150 mg once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22.
- TMC435 200 mg (Cohort 4/Panel C): Treatment-experienced non-responders received TMC435 200 mg once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22.
- Placebo (Cohort 4/Panel C): Treatment-experienced non-responders received placebo (identical in appearance to TMC435 75 mg, 150 mg, or 200 mg) once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22.
- TMC435 200 mg (Cohort 5/Panel D): Treatment-experienced relapsers received TMC435 200 mg once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22.
Period: Overall Study
Arm/Group | TMC435 25 mg (Cohort 1/Panel A and B) | TMC435 75mg (Cohort 1/Panel A and B) | Placebo (Cohort 1/Panel A and B) | TMC435 200 mg (Cohort 2, Panel A and B) | Placebo (Cohort 2/Panel A and B) | TMC435 75 mg (Cohort 4/Panel C) | TMC435 150 mg (Cohort 4/Panel C) | TMC435 200 mg (Cohort 4/Panel C) | Placebo (Cohort 4/Panel C) | TMC435 200 mg (Cohort 5/Panel D)
Started | 18 | 19 | 13 | 18 | 6 | 9 | 9 | 10 | 9 | 5
Completed | 13 | 16 | 10 | 12 | 5 | 3 | 3 | 6 | 2 | 3
Not Completed | 5 | 3 | 3 | 6 | 1 | 6 | 6 | 4 | 7 | 2
Not completed — Subject reached a virologic endpoint | 2 | 1 | 1 | 4 | 1 | 3 | 4 | 4 | 5 | 0
Not completed — Subject ineligible to continue the trial | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 1
Not completed — Other | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Lost to Follow-up | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- TMC435 25 mg (Cohort 1): Treatment-naïve participants received TMC435 25 mg once daily for 7 days followed by TMC435 25 mg once daily coadministered with ribavirin (RBV) for 21 days + peginterferon alpha-2a (PegIFNα-2a) on Days 8, 15, and 22 (Panel A) OR TMC435 25 mg once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22 (Panel B)
- TMC435 75mg (Cohort 1): Treatment-naïve participants received TMC435 75 mg once daily for 7 days followed by TMC435 75 mg once daily coadministered with RBV for 21 days + PegIFNα-2a on Days 8, 15, and 22 (Panel A) OR TMC435 75 mg once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22 (Panel B)
- Placebo (Cohort 1): Treatment-naïve participants received placebo (identical in appearance to TMC435 25 mg or 75 mg) once daily for 7 days followed by placebo once daily coadministered with RBV for 21 days + PegIFNα-2a on Days 8, 15, and 22 (Panel A) OR placebo once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22 (Panel B)
- TMC435 200 mg (Cohort 2): Treatment-naïve participants received TMC435 200 mg once daily for 7 days followed by TMC435 200 mg once daily coadministered with RBV for 21 days + PegIFNα-2a on Days 8, 15, and 22 (Panel A) OR TMC435 200 mg once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22 (Panel B)
- Placebo (Cohort 2): Treatment-naïve participants received placebo (identical in appearance to TMC435 200 mg) once daily for 7 days followed by placebo once daily coadministered with RBV for 21 days + PegIFNα-2a on Days 8, 15, and 22 (Panel A) OR placebo once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22 (Panel B)
- TMC435 75 mg (Cohort 4): Treatment-experienced non-responders received TMC435 75 mg once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22.
- TMC435 150 mg (Cohort 4): Treatment-experienced non-responders received TMC435 150 mg once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22.
- TMC435 200 mg (Cohort 4): Treatment-experienced non-responders received TMC435 200 mg once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22.
- Placebo (Cohort 4): Treatment-experienced non-responders received placebo (identical in appearance to TMC435 75 mg, 150 mg, or 200 mg) once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22.
- TMC435 200 mg (Cohort 5): Treatment-experienced relapsers received TMC435 200 mg once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22.
- Total: Total of all reporting groups
Arm/Group | TMC435 25 mg (Cohort 1) | TMC435 75mg (Cohort 1) | Placebo (Cohort 1) | TMC435 200 mg (Cohort 2) | Placebo (Cohort 2) | TMC435 75 mg (Cohort 4) | TMC435 150 mg (Cohort 4) | TMC435 200 mg (Cohort 4) | Placebo (Cohort 4) | TMC435 200 mg (Cohort 5) | Total
Number analyzed (Participants) | 18 | 19 | 13 | 18 | 6 | 9 | 9 | 10 | 9 | 5 | 116
Age, Continuous [Median (Full Range); unit: years] | 52 [22 to 64] | 47 [22 to 70] | 45 [19 to 60] | 46.5 [19 to 68] | 44.5 [19 to 50] | 53 [38 to 62] | 56 [32 to 67] | 55.5 [28 to 69] | 47 [21 to 57] | 56 [33 to 66] | 49 [19 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 3 | 8 | 1 | 3 | 1 | 2 | 0 | 0 | 31
  Male | 13 | 11 | 10 | 10 | 5 | 6 | 8 | 8 | 9 | 5 | 85
The Number of Participants Randomized to each Treatment Panel [Number; unit: participants] — The table below shows the number of participants in Cohorts 1, 2, 4 and 5 that were randomized to treatment Panels A, B, C, and D.
  participants
    Panel A | 9 | 10 | 6 | 9 | 3 | 0 | 0 | 0 | 0 | 0 | 37
    Panel B | 9 | 9 | 7 | 9 | 3 | 0 | 0 | 0 | 0 | 0 | 37
    Panel C | 0 | 0 | 0 | 0 | 0 | 9 | 9 | 10 | 9 | 0 | 37
    Panel D | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Plasma Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Levels (log10 IU/mL) at Week 4 in Treatment-Naïve HCV-Infected Participants (Cohort 1 and 2, Panel A)
Description: The table below shows the change from Baseline in plasma levels of HCV RNA at Week 4 following treatment with TMC435 or placebo as for 7 days followed by TMC435 or placebo coadministered with ribavirin for 21 days + peginterferon alpha-2a (PegIFNα-2a) on Days 1, 8, 15, and 22 in treatment-naïve HCV-infected participants. (A treatment-naive participant is someone who has never taken drugs for their HCV infection).
Time Frame: Week 4
Population: The intent-to-treat population (defined as all participants who were randomized and received at least one dose of study medication) was used for all analyses.
Measure: Mean (Standard Error); unit: log10 IU/mL
Groups:
- TMC435 25 mg (Cohort 1, Panel A): Treatment-naïve participants received TMC435 25 mg once daily for 7 days followed by TMC435 25 mg once daily coadministered with ribavirin (RBV) for 21 days + peginterferon alpha-2a (PegIFNα-2a) on Days 8, 15, and 22.
- TMC435 75 mg (Cohort 1, Panel A): Treatment-naïve participants received TMC435 75 mg once daily for 7 days followed by TMC435 75 mg once daily coadministered with RBV for 21 days + PegIFNα-2a on Days 8, 15, and 22.
- Placebo (Cohort 1, Panel A): Treatment-naïve participants received placebo (identical in appearance to TMC435 25 or 75 mg) once daily for 7 days followed by placebo once daily coadministered with RBV for 21 days + PegIFNα-2a on Days 8, 15, and 22.
- TMC435 200 mg (Cohort 2, Panel A): Treatment-naïve participants received TMC435 200 mg once daily for 7 days followed by TMC435 200 mg once daily coadministered with RBV for 21 days + PegIFNα-2a on Days 8, 15, and 22.
- Placebo (Cohort 2, Panel A): Treatment-naïve participants received placebo (identical in appearance to TMC435 200 mg) once daily for 7 days followed by placebo once daily coadministered with RBV for 21 days + PegIFNα-2a on Days 8, 15, and 22.
Arm/Group | TMC435 25 mg (Cohort 1, Panel A) | TMC435 75 mg (Cohort 1, Panel A) | Placebo (Cohort 1, Panel A) | TMC435 200 mg (Cohort 2, Panel A) | Placebo (Cohort 2, Panel A)
Number analyzed (Participants) | 9 | 10 | 6 | 9 | 3
log10 IU/mL | -4.26 (0.646) | -4.47 (0.489) | -2.97 (0.640) | -4.70 (0.584) | -1.92 (0.156)

2. Primary Outcome: Change From Baseline in Plasma Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Levels (log10 IU/mL) at Week 4 in Treatment-Naïve HCV-Infected Participants (Cohort 1 and 2, Panel B)
Description: The table below shows the change from Baseline in plasma levels of HCV RNA at Week 4 following treatment with TMC435 or placebo coadministered with ribavirin for 28 days + peginterferon alpha-2a (PegIFNα-2a) on Days 1, 8, 15, and 22 in treatment-naïve HCV-infected participants. (A treatment-naive participant is someone who has never taken drugs for their HCV infection).
Time Frame: Week 4
Population: as for outcome 1
Measure: Mean (Standard Error); unit: log10 IU/mL
Groups:
- TMC435 25 mg (Cohort 1, Panel B): Treatment-naïve participants received TMC435 25 mg once daily coadministered with ribavirin (RBV) for 28 days + peginterferon alpha-2a (PegIFNα-2a) on Days 1, 8, 15, and 22.
- TMC435 75 mg (Cohort 1, Panel B): Treatment-naïve participants received TMC435 75 mg once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22.
- Placebo (Cohort 1, Panel B): Treatment-naïve participants received placebo (identical in appearance to TMC435 25 mg or 75 mg) once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22.
- TMC435 200 mg (Cohort 2, Panel B): Treatment-naïve participants received TMC435 200 mg once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22.
- Placebo (Cohort 2, Panel B): Treatment-naïve participants received placebo (identical in appearance to TMC435 200 mg) once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22.
Arm/Group | TMC435 25 mg (Cohort 1, Panel B) | TMC435 75 mg (Cohort 1, Panel B) | Placebo (Cohort 1, Panel B) | TMC435 200 mg (Cohort 2, Panel B) | Placebo (Cohort 2, Panel B)
Number analyzed (Participants) | 9 | 9 | 7 | 9 | 3
log10 IU/mL | -4.74 (0.455) | -5.52 (0.228) | -3.74 (0.665) | -5.44 (0.169) | -3.26 (1.222)

3. Primary Outcome: Change From Baseline in Plasma Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Levels (log10 IU/mL) at Week 4 in Treatment-Experienced HCV-Infected Participants (Cohort 4, Panel C and Cohort 5, Panel D)
Description: The table below shows the change from Baseline in plasma levels of HCV RNA at Week 4 following treatment with TMC435 or placebo coadministered with ribavirin for 28 days + peginterferon alpha-2a (PegIFNα-2a) on Days 1, 8, 15, and 22 in treatment-experienced participants considered non-responders (defined as participants who achieved less than a 2 log10 IU/mL decline from baseline in plasma HCV RNA levels after 12 weeks of previous interferon [IFN]-based therapy [pegylated or non-pegylated]) or relapsers (defined as a participant with undetectable plasma HCV RNA at the end of treatment of previous IFN-based therapy and subsequent confirmed detectable plasma HCV RNA levels during follow-up).
Time Frame: Week 4
Population: as for outcome 1
Measure: Mean (Standard Error); unit: log10 IU/mL
Groups:
- TMC435 75 mg (Cohort 4, Panel C): Treatment-experienced non-responders received TMC435 75 mg once daily coadministered with ribavirin (RBV) for 28 days + peginterferon alpha-2a (PegIFNα-2a) on Days 1, 8, 15, and 22.
- TMC435 150 mg (Cohort 4, Panel C): Treatment-experienced non-responders received TMC435 150 mg once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22.
- TMC435 200 mg (Cohort 4, Panel C): Treatment-experienced non-responders received TMC435 200 mg once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22.
- Placebo (Cohort 4, Panel C): Treatment-experienced non-responders received placebo (identical in appearance to TMC435 75 mg, 150 mg, or 200 mg) once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22.
- TMC435 200 mg (Cohort 5, Panel D): Treatment-experienced relapsers received TMC435 200 mg once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22.
Arm/Group | TMC435 75 mg (Cohort 4, Panel C) | TMC435 150 mg (Cohort 4, Panel C) | TMC435 200 mg (Cohort 4, Panel C) | Placebo (Cohort 4, Panel C) | TMC435 200 mg (Cohort 5, Panel D)
Number analyzed (Participants) | 9 | 9 | 10 | 9 | 4
log10 IU/mL | -4.28 (0.539) | -5.46 (0.425) | -5.26 (0.238) | -1.53 (0.216) | -5.86 (0.198)

4. Secondary Outcome: Change From Baseline in Plasma Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Levels (log10 IU/mL) on Day 7 in Treatment-Naïve HCV-Infected Participants (Cohort 1 and 2, Panel A)
Description: The table below shows the change from Baseline in plasma levels of HCV RNA on Day 7 (at Week 1) following treatment with TMC435 or placebo for 7 days followed by TMC435 or placebo coadministered with ribavirin for 21 days + peginterferon alpha-2a (PegIFNα-2a) on Days 8, 15, and 22 in treatment-naïve HCV-infected participants. (A treatment-naive participant is someone who has never taken drugs for their HCV infection).
Time Frame: Day 7
Population: as for outcome 1
Measure: Mean (Standard Error); unit: log10 IU/mL
Groups:
- Placebo (Cohort 2, Panel A): Treatment-naïve participants in received placebo (identical in appearance to TMC435 200 mg) once daily for 7 days followed by placebo once daily coadministered with RBV for 21 days + PegIFNα-2a on Days 8, 15, and 22.
Arm/Group | TMC435 25 mg (Cohort 1, Panel A) | TMC435 75 mg (Cohort 1, Panel A) | Placebo (Cohort 1, Panel A) | TMC435 200 mg (Cohort 2, Panel A) | Placebo (Cohort 2, Panel A)
Number analyzed (Participants) | 9 | 10 | 6 | 9 | 3
log10 IU/mL | -2.63 (0.377) | -3.48 (0.285) | -0.08 (0.101) | -4.18 (0.158) | 0.30 (0.080)

5. Secondary Outcome: Change From Baseline in Plasma Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Levels (log10 IU/mL) on Day 7 in Treatment-Naïve HCV-Infected Participants (Cohort 1 and 2, Panel B)
Description: The table below shows the change from Baseline in plasma levels of HCV RNA on Day 7 (at Week 1) following treatment with TMC435 or placebo coadministered with ribavirin for 28 days + peginterferon alpha-2a (PegIFNα-2a) on Days 1, 8, 15, and 22 in treatment-naïve HCV-infected participants (A treatment-naive participant is someone who has never taken drugs for their HCV infection).
Time Frame: Day 7
Population: as for outcome 1
Measure: Mean (Standard Error); unit: log10 IU/mL
Groups:
- TMC435 200 mg (Cohort 2, Panel B): Treatment-naïve participants received TMC435 200 mg once daily for 28 days coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22.
Arm/Group | TMC435 25 mg (Cohort 1, Panel B) | TMC435 75 mg (Cohort 1, Panel B) | Placebo (Cohort 1, Panel B) | TMC435 200 mg (Cohort 2, Panel B) | Placebo (Cohort 2, Panel B)
Number analyzed (Participants) | 9 | 9 | 7 | 9 | 3
log10 IU/mL | -3.47 (0.500) | -4.55 (0.192) | -1.73 (0.441) | -4.68 (0.135) | -1.64 (0.793)

6. Secondary Outcome: Change From Baseline in Plasma Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Levels (log10 IU/mL) on Day 7 in Treatment-Experienced HCV-Infected Participants (Cohort 4, Panel C and Cohort 5, Panel D)
Description: The table below shows the change from Baseline in plasma levels of HCV RNA on Day 7 (Week 1) following treatment with TMC435 or placebo coadministered with ribavirin for 28 days + peginterferon alpha-2a (PegIFNα-2a) on Days 1, 8, 15, and 22 in treatment-experienced participants considered non-responders (defined as participants who achieved less than a 2 log10 IU/mL decline from baseline in plasma HCV RNA levels after 12 weeks of previous interferon [IFN]-based therapy [pegylated or non-pegylated]) or relapsers (defined as a participant with undetectable plasma HCV RNA at the end of treatment of previous IFN-based therapy and subsequent confirmed detectable plasma HCV RNA levels during follow-up).
Time Frame: Day 7
Population: as for outcome 1
Measure: Mean (Standard Error); unit: log10 IU/mL
Arm/Group | TMC435 75 mg (Cohort 4, Panel C) | TMC435 150 mg (Cohort 4, Panel C) | TMC435 200 mg (Cohort 4, Panel C) | Placebo (Cohort 4, Panel C) | TMC435 200 mg (Cohort 5, Panel D)
Number analyzed (Participants) | 9 | 9 | 10 | 9 | 5
log10 IU/mL | -3.80 (0.432) | -4.68 (0.224) | -4.49 (0.318) | -0.50 (0.152) | -4.08 (0.387)

7. Secondary Outcome: Virologic Responses Following Treatment With TMC435 in Treatment-Naive Hepatitis C Virus (HCV)-Infected Participants (Cohort 1 and 2, Panel A)
Description: The table below shows the number of treatment-naïve HCV-infected participants treated with TMC435 or placebo for 7 days followed by TMC435 or placebo coadministered with ribavirin for 21 days + peginterferon alpha-2a (PegIFNα-2a) on Days 8, 15, and 22 who had the following virologic responses: plasma levels of HCV ribonucleic acid (RNA) of greater than or equal to 2 log10 decline from Baseline; plasma levels of HCV RNA below the limit of quantification (ie, less than [<] 25 IU/mL detectable or undetectable); plasma levels of HCV RNA below the limit of detection (ie, <25 IU/mL undetectable); plasma levels of HCV RNA <100 IU/mL; and plasma levels of HCV RNA <1000 at the time points listed. See "treatment-naive" defined above.
Time Frame: Day 2 or 3, Day 7, and Day 28
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | TMC435 25 mg (Cohort 1, Panel A) | TMC435 75 mg (Cohort 1, Panel A) | Placebo (Cohort 1, Panel A) | TMC435 200 mg (Cohort 2, Panel A) | Placebo (Cohort 2, Panel A)
Number analyzed (Participants) | 9 | 10 | 6 | 9 | 3
Participants
  Day 2/3: > or = 2 log10 change from baseline | 6 (0.646) | 9 (0.489) | 0 (0.640) | 9 (0.584) | 0 (0.156)
  Day 7: > or = 2 log10 change from baseline | 7 | 9 | 0 | 9 | 0
  Day 28: > or = 2 log10 change from baseline | 7 | 9 | 4 | 8 | 1
  Day 2/3: <25 IU/mL detectable or undetectable | 1 | 1 | 0 | 1 | 0
  Day 7: <25 IU/mL detectable or undetectable | 1 | 0 | 0 | 1 | 0
  Day 28: <25 IU/mL detectable or undetectable | 5 | 8 | 1 | 7 | 0
  Day 2/3: <25 IU/mL undetectable | 0 | 0 | 0 | 0 | 0
  Day 7: <25 IU/mL undetectable | 0 | 0 | 0 | 0 | 0
  Day 28: <25 IU/mL undetectable | 5 | 5 | 1 | 7 | 0
  Day 2/3: <100 IU/mL | 1 | 1 | 0 | 1 | 0
  Day 7: <100 IU/mL | 1 | 3 | 0 | 4 | 0
  Day 28: <100 IU/mL | 6 | 8 | 1 | 7 | 0
  Day 2/3: <1000 IU/mL | 2 | 5 | 0 | 6 | 0
  Day 7: <1000 IU/mL | 3 | 6 | 0 | 7 | 0
  Day 28: <1000 IU/mL | 7 | 8 | 2 | 7 | 0

8. Secondary Outcome: Virologic Responses Following Treatment With TMC435 in Treatment-Naive Hepatitis C Virus (HCV)-Infected Participants (Cohort 1 and 2, Panel B)
Description: The table below shows the number of treatment-naive HCV-Infected participants with the following virologic responses to treatment with TMC435 or placebo coadministered with ribavirin for 28 days + peginterferon alpha-2a (PegIFNα-2a) on Days 8, 15, and 22: plasma levels of HCV ribonucleic acid (RNA) of greater than or equal to 2 log10 decline from Baseline; plasma levels of HCV RNA below the limit of quantification (ie, less than [<] 25 IU/mL detectable or undetectable); plasma levels of HCV RNA below the limit of detection (ie, <25 IU/mL undetectable); plasma levels of HCV RNA <100 IU/mL; and plasma levels of HCV RNA <1000 at the time points listed. See "treatment-naive" defined above.
Time Frame: Day 2 or 3, Day 7, and Day 28
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- TMC435 25 (Cohort 1, Panel B): Treatment-naïve participants received TMC435 25 mg once daily coadministered with ribavirin (RBV) for 28 days + peginterferon alpha-2a (PegIFNα-2a) on Days 1, 8, 15, and 22.
- Placebo (Cohort 1, Panel B): Treatment-naïve participants received placebo (identical in appearance to TMC435 25 mg and 75 mg) once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22.
Arm/Group | TMC435 25 (Cohort 1, Panel B) | TMC435 75 mg (Cohort 1, Panel B) | Placebo (Cohort 1, Panel B) | TMC435 200 mg (Cohort 2, Panel B) | Placebo (Cohort 2, Panel B)
Number analyzed (Participants) | 9 | 9 | 7 | 9 | 3
Participants
  Day 2/3: > or = 2 log10 change from baseline | 7 (0.646) | 9 (0.489) | 2 (0.640) | 9 (0.584) | 2 (0.156)
  Day 7: > or = 2 log10 change from baseline | 7 | 9 | 2 | 9 | 1
  Day 28: > or = 2 log10 change from baseline | 8 | 9 | 6 | 9 | 2
  Day 2/3: <25 IU/mL detectable or undetectable | 0 | 0 | 0 | 0 | 0
  Day 7: <25 IU/mL detectable or undetectable | 1 | 1 | 0 | 3 | 0
  Day 28: <25 IU/mL detectable or undetectable | 6 | 9 | 3 | 9 | 1
  Day 2/3: <25 IU/mL undetectable | 0 | 0 | 0 | 0 | 0
  Day 7: <25 IU/mL undetectable | 0 | 0 | 0 | 1 | 0
  Day 28: <25 IU/mL undetectable | 3 | 8 | 2 | 6 | 0
  Day 2/3: <100 IU/mL | 0 | 1 | 0 | 1 | 0
  Day 7: <100 IU/mL | 1 | 6 | 0 | 5 | 0
  Day 28: <100 IU/mL | 6 | 9 | 3 | 9 | 1
  Day 2/3: <1000 IU/mL | 4 | 5 | 0 | 6 | 0
  Day 7: <1000 IU/mL | 5 | 9 | 0 | 9 | 0
  Day 28: <1000 IU/mL | 7 | 9 | 4 | 9 | 2

9. Secondary Outcome: Virologic Responses Following Treatment With TMC435 in Treatment-Experienced Hepatitis C Virus (HCV)-Infected Participants (Cohort 4, Panel C and Cohort 5, Panel D)
Description: The table below shows the number of treatment-experienced participants (non-responders and relapsers, see defined above) with the following virologic responses to treatment with TMC435 or placebo coadministered with ribavirin for 28 days + peginterferon alpha-2a (PegIFNα-2a) on Days 1, 8, 15, and 22: plasma levels of HCV ribonucleic acid (RNA) of greater than or equal to 2 log10 decline from Baseline; plasma levels of HCV RNA below the limit of quantification (ie, less than [<] 25 IU/mL detectable or undetectable); plasma levels of HCV RNA below the limit of detection (ie, <25 IU/mL undetectable); plasma levels of HCV RNA <100 IU/mL; and plasma levels of HCV RNA <1000 at the time points listed. Note: in the table below, the number of participants (n) analyzed in the TMC435 200 mg (Cohort 4, Panel B) on Day 28 (Week 4) was n=4.
Time Frame: Day 2 or 3, Day 7, and Day 28
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | TMC435 75 mg (Cohort 4, Panel C) | TMC435 150 mg (Cohort 4, Panel C) | TMC435 200 mg (Cohort 4, Panel C) | Placebo (Cohort 4, Panel C) | TMC435 200 mg (Cohort 5, Panel D)
Number analyzed (Participants) | 9 | 9 | 10 | 9 | 5
Participants
  Day 2/3: > or = 2 log10 change from baseline | 8 (0.646) | 9 (0.489) | 10 (0.640) | 1 (0.584) | 4 (0.156)
  Day 7: > or = 2 log10 change from baseline | 8 | 9 | 10 | 0 | 5
  Day 28: > or = 2 log10 change from baseline | 8 | 9 | 10 | 2 | 4
  Day 2/3: <25 IU/mL detectable or undetectable | 0 | 0 | 0 | 0 | 0
  Day 7: <25 IU/mL detectable or undetectable | 0 | 2 | 3 | 0 | 0
  Day 28: <25 IU/mL detectable or undetectable | 4 | 7 | 7 | 0 | 4
  Day 2/3: <25 IU/mL undetectable | 0 | 0 | 0 | 0 | 0
  Day 7: <25 IU/mL undetectable | 0 | 0 | 0 | 0 | 0
  Day 28: <25 IU/mL undetectable | 2 | 5 | 3 | 0 | 3
  Day 2/3: <100 IU/mL | 0 | 0 | 0 | 0 | 0
  Day 7: <100 IU/mL | 2 | 4 | 5 | 0 | 0
  Day 28: <100 IU/mL | 6 | 8 | 7 | 0 | 4
  Day 2/3: <1000 IU/mL | 3 | 3 | 5 | 0 | 0
  Day 7: <1000 IU/mL | 5 | 7 | 8 | 0 | 3
  Day 28: <1000 IU/mL | 6 | 8 | 10 | 0 | 4

10. Secondary Outcome: Virologic Response Parameters in Treatment-Naïve Hepatitis C Virus (HCV)-Infected Participants (Cohort 1 and 2, Panel A and B Combined)
Description: The table below shows the number of treatment-naïve participants in the treatment groups for Cohort 1 (Panel A and B combined) and in Cohort 2 (Panel A and B combined) who met the following virologic response parameters: rapid virological response (RVR) defined as having undetectable plasma HCV ribonucleic acid (RNA) at Week 4; early virologic response (EVR) defined as change from baseline in plasma HCV RNA of greater than or equal to 2 log 10 at Week 12); a complete EVR (cEVR) defined as a complete EVR having undetectable plasma HCV RNA at Week 12); an extended RVR (eRVR) defined as undetectable plasma HCV RNA at Week 4 and 12; and a partial response defined as EVR but not reaching undetectability while on treatment.
Time Frame: Week 4 (RVR), Week 12 (EVR, cEVR, and partial response), and Week 4 and 12 (eRVR)
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- TMC435 25 mg (Cohort 1, Panel A and B): Treatment-naïve participants received TMC435 25 mg once daily for 7 days followed by TMC435 25 mg once daily coadministered with ribavirin (RBV) for 21 days + peginterferon alpha-2a (PegIFNα-2a) on Days 8, 15, and 22 (Panel A) OR TMC435 25 mg once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22 (Panel B).
- TMC435 75mg (Cohort 1, Panel A and B): Treatment-naïve participants received TMC435 75 mg once daily for 7 days followed by TMC435 25 mg once daily coadministered with RBV for 21 days + PegIFNα-2a on Days 8, 15, and 22 (Panel A) OR TMC435 75 mg once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22 (Panel B).
- Placebo (Cohort 1, Panel A and B): Treatment-naïve participants received placebo (identical in appearance to TMC435 25 mg or 75 mg) once daily for 7 days followed RBV for 21 days + PegIFNα-2a on Days 8, 15, and 22 (Panel A) OR placebo once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22 (Panel B).
- TMC435 200mg (Cohort 2, Panel A and B): Treatment-naïve participants received TMC435 200 mg once daily for 7 days followed by TMC435 200 mg once daily coadministered with RBV for 21 days + PegIFNα-2a on Days 8, 15, and 22 (Panel A) OR TMC435 200 mg once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22 (Panel B).
- Placebo (Cohort 2, Panel A and B): Treatment-naïve participants received placebo (identical in appearance to TMC435 200 mg) once daily for 7 days followed RBV for 21 days + PegIFNα-2a on Days 8, 15, and 22 (Panel A) OR placebo once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22 (Panel B).
Arm/Group | TMC435 25 mg (Cohort 1, Panel A and B) | TMC435 75mg (Cohort 1, Panel A and B) | Placebo (Cohort 1, Panel A and B) | TMC435 200mg (Cohort 2, Panel A and B) | Placebo (Cohort 2, Panel A and B)
Number analyzed (Participants) | 18 | 19 | 13 | 18 | 6
Participants
  RVR | 8 (0.646) | 13 (0.489) | 3 (0.640) | 13 (0.584) | 0 (0.156)
  EVR | 16 | 19 | 12 | 16 | 6
  cEVR | 13 | 17 | 7 | 16 | 5
  eRVR | 8 | 13 | 3 | 13 | 0
  Partial response | 0 | 0 | 0 | 0 | 1

11. Secondary Outcome: Virologic Response Parameters Following Treatment With TMC435 in Treatment-Experienced Hepatitis C Virus (HCV)-Infected Participants (Cohort 4, Panel C and Cohort 5, Panel D)
Description: The table below shows the number of treatment-experienced participants (non-responders and relapsers, see defined above) treated with TMC435 or placebo coadministered with ribavirin for 28 days + peginterferon alpha-2a (PegIFNα-2a) on Days 1, 8, 15, and 22 who met the following virologic response parameters: rapid virological response (RVR) defined as having undetectable plasma HCV ribonucleic acid (RNA) at Week 4; early virologic response (EVR) defined as change from baseline in plasma HCV RNA of greater than or equal to 2 log 10 at Week 12; a complete EVR (cEVR) defined as a EVR having undetectable plasma HCV RNA at Week 12; an extended RVR (eRVR) defined as undetectable plasma HCV RNA at Week 4 and 12; and a partial response defined as EVR but not reaching undetectability while on treatment.
Time Frame: Week 4 (RVR), Week 12 (EVR, cEVR, and partial response), and Week 4 and 12 (eRVR)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | TMC435 75 mg (Cohort 4, Panel C) | TMC435 150 mg (Cohort 4, Panel C) | TMC435 200 mg (Cohort 4, Panel C) | Placebo (Cohort 4, Panel C) | TMC435 200 mg (Cohort 5, Panel D)
Number analyzed (Participants) | 9 | 9 | 10 | 9 | 5
Participants
  RVR | 2 (0.646) | 5 (0.489) | 3 (0.640) | 0 (0.584) | 3 (0.156)
  EVR | 6 | 7 | 8 | 8 | 4
  cEVR | 4 | 4 | 5 | 0 | 3
  eRVR | 2 | 4 | 3 | 0 | 3
  Partial response | 0 | 1 | 1 | 5 | 0

12. Secondary Outcome: Initial Suboptimal Responses Following Treatment With TMC435 in Treatment-Naïve Hepatitis C Virus (HCV)-Infected Participants (Cohort 1 and 2, Panel A)
Description: The table below shows the number of treatment-naïve participants with an initial suboptimal response defined as less than 2 log10 change in plasma level of hepatitis C virus (HCV) ribonucleic acid (RNA) on Day 2 or 3 (depending when visit was scheduled) following treatment with TMC435 or placebo for 7 days followed by TMC435 or placebo coadministered with ribavirin for 21 days + peginterferon alpha-2a (PegIFNα-2a) on Days 8, 15, and 22. See "treatment-naive" defined above.
Time Frame: Day 2 or 3
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- Placebo (Cohort 1, Panel A): Treatment-naïve participants received placebo identical in appearance toTMC435 25 or 75 mg) once daily for 7 days followed by placebo once daily coadministered with RBV for 21 days + PegIFNα-2a on Days 8, 15, and 22.
Arm/Group | TMC435 25 mg (Cohort 1, Panel A) | TMC435 75 mg (Cohort 1, Panel A) | Placebo (Cohort 1, Panel A) | TMC435 200 mg (Cohort 2, Panel A) | Placebo (Cohort 2, Panel A)
Number analyzed (Participants) | 9 | 10 | 6 | 9 | 3
Participants | 3 | 1 | 6 | 0 | 3

13. Secondary Outcome: Initial Suboptimal Responses Following Treatment With TMC435 in Treatment-Naïve Hepatitis C Virus (HCV)-Infected Participants (Cohort 1 and 2, Panel B)
Description: The table below shows the number of treatment-naïve participants with an initial suboptimal response defined as less than 2 log10 change in plasma plasma level of hepatitis C virus (HCV) ribonucleic acid (RNA) on Day 2 or 3 (depending when visit was scheduled) after treatment with TMC435 or placebo coadministered with ribavirin for 28 days + peginterferon alpha-2a (PegIFNα-2a) on Days 1, 8, 15, and 22. See "treatment-naive" defined above.
Time Frame: Day 2 or 3
Population: The intent-to-treat (ITT) population, defined as all participants who were randomized and received at least one dose of study medication (TMC435) was used for all analyses.
Measure: Number; unit: Participants
Groups:
- TMC435 25 mg (Cohort 1, Panel B): Treatment-naïve participants received TMC435 25 mg coadministered with ribavirin (RBV) for 28 days + peginterferon alpha-2a (PegIFNα-2a) on Days 1, 8, 15, and 22.
- TMC435 75 mg (Cohort 1, Panel B): Treatment-naïve participants received TMC435 75 mg once daily for 28 days coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22.
Arm/Group | TMC435 25 mg (Cohort 1, Panel B) | TMC435 75 mg (Cohort 1, Panel B) | Placebo (Cohort 1, Panel B) | TMC435 200 mg (Cohort 2, Panel B) | Placebo (Cohort 2, Panel B)
Number analyzed (Participants) | 9 | 9 | 7 | 9 | 3
Participants | 2 (0.646) | 0 (0.489) | 5 (0.640) | 0 (0.584) | 1 (0.156)

14. Secondary Outcome: Initial Suboptimal Responses Following Treatment With TMC435 in Treatment-Experienced Hepatitis C Virus (HCV)-Infected Participants (Cohort 4, Panel C and Cohort 5, Panel D)
Description: The table below shows the number of treatment-experienced participants (non-responders and relapsers, see defined above) with an initial suboptimal response defined as less than 2 log10 change of plasma in plasma level of HCV ribonucleic acid (RNA) at Day 2 or 3 (depending when visit was scheduled) treated with TMC435 or placebo coadministered with ribavirin for 28 days + peginterferon alpha-2a (PegIFNα-2a) on Days 1, 8, 15, and 22.
Time Frame: Day 2 or 3
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | TMC435 75 mg (Cohort 4, Panel C) | TMC435 150 mg (Cohort 4, Panel C) | TMC435 200 mg (Cohort 4, Panel C) | Placebo (Cohort 4, Panel C) | TMC435 200 mg (Cohort 5, Panel D)
Number analyzed (Participants) | 9 | 9 | 10 | 9 | 5
Participants | 1 | 0 | 0 | 8 | 1

15. Secondary Outcome: Viral Breakthrough in Treatment-Naïve Hepatitis C Virus (HCV)-Infected Participants (Cohort 1, Panel A and B)
Description: The table below shows the number of treatment-naïve participants with viral breakthrough, defined as a confirmed increase of greater than 1 log10 IU/mL in plasma HCV ribonucleic acid (RNA) level from the lowest level reached, or a confirmed plasma HCV RNA level of greater than 100 IU/mL in participants whose plasma HCV RNA had previously been below the limit of quantification (25 IU/mL detectable) or undetectable (less than 25 IU/mL undetectable) after treatment with TMC435 or placebo for 7 days followed by TMC435 or placebo coadministered with ribavirin for 21 days + peginterferon alpha-2a (PegIFNα-2a) on days 8, 15, and 22 (Panel A) and after treatment with TMC435 or placebo coadministered with ribavirin for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22 (Panel B).
Time Frame: 4 Weeks (Wks), 44 Wks, and 48 Wks
Population: The intent-to-treat population (defined as all participants who were randomized and received at least one dose of study medication) was used for all analyses. Note: Number of participants analyzed during the PegIFNα-2a and ribavirin treatment period of up to 44 weeks is N=16 for TMC435 25 mg, N=17 for TMC435 75 mg, and N=17 for TMC435 200 mg.
Measure: Number; unit: Participants
Groups:
- TMC435 25 mg (Cohort 1, Panels A and B): Treatment-naïve participants received TMC435 25 mg once daily for 7 days followed by TMC435 25 mg once daily coadministered with ribavirin (RBV) for 21 days + peginterferon alpha-2a (PegIFNα-2a) on Days 8, 15, and 22 (Panel A) OR TMC435 25 mg once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22 (Panel B).
- TMC435 75 mg (Cohort 1, Panels A and B): Treatment-naïve participants received TMC435 75 mg once daily for 7 days followed by TMC435 25 mg once daily coadministered with RBV for 21 days + PegIFNα-2a on Days 8, 15, and 22 (Panel A) OR TMC435 75 mg once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22 (Panel B).
- Placebo (Cohort 1, Panels A and B): Treatment-naïve participants received placebo (identical in appearance to TMC435 25 mg or 75 mg) once daily for 7 days followed RBV for 21 days + PegIFNα-2a on Days 8, 15, and 22 (Panel A) OR placebo once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22 (Panel B).
- TMC435 200 mg (Cohort 2, Panels A and B): Treatment-naïve participants received TMC435 200 mg once daily for 7 days followed by TMC435 200 mg once daily coadministered with RBV for 21 days + PegIFNα-2a on Days 8, 15, and 22 (Panel A) OR TMC435 200 mg once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22 (Panel B).
- Placebo (Cohort 2, Panels A and B): Treatment-naïve participants received placebo (identical in appearance to TMC435 200 mg) once daily for 7 days followed RBV for 21 days + PegIFNα-2a on Days 8, 15, and 22 (Panel A) OR placebo once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22 (Panel B).
Arm/Group | TMC435 25 mg (Cohort 1, Panels A and B) | TMC435 75 mg (Cohort 1, Panels A and B) | Placebo (Cohort 1, Panels A and B) | TMC435 200 mg (Cohort 2, Panels A and B) | Placebo (Cohort 2, Panels A and B)
Number analyzed (Participants) | 18 | 19 | 13 | 18 | 6
Participants
  Entire treatment period (48 Wks) | 3 | 3 | 0 | 4 | 0
  During TMC435/Placebo treatment (4 Wks) | 2 | 2 | 0 | 1 | 0
  During treatment with RBV and PegIFNα-2a (44 Wks) | 1 | 1 | 0 | 3 | 0

16. Secondary Outcome: Viral Breakthrough in Treatment-Experienced Hepatitis C Virus (HCV)-Infected Participants (Cohort 4, Panel C and Cohort 5, Panel D)
Description: The table below shows the number of treatment-experienced participants (non-responders and relapsers, see defined above) with viral breakthrough, defined as a confirmed increase of greater than 1 log10 IU/mL in plasma HCV ribonucleic acid (RNA) level from the lowest level reached), or a confirmed plasma HCV RNA level of greater than 100 IU/mL in participants whose plasma HCV RNA had previously been below the limit of quantification (25 IU/mL detectable) or undetectable (less than 25 IU/mL undetectable) treated with TMC435 or placebo coadministered with ribavirin for 28 days + peginterferon alpha-2a (PegIFNα-2a) on Days 1, 8, 15, and 22.
Time Frame: 4 Weeks (Wks), 44 Wks, and 48 Wks
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- Placebo (TMC435 75/150/200 mg) (Cohort 4, Panel C): Treatment-experienced non-responders received Placebo identical in appearance to TMC435 75 mg, 150 mg, or 200 mg once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22.
Arm/Group | TMC435 75 mg (Cohort 4, Panel C) | TMC435 150 mg (Cohort 4, Panel C) | TMC435 200 mg (Cohort 4, Panel C) | Placebo (TMC435 75/150/200 mg) (Cohort 4, Panel C) | TMC435 200 mg (Cohort 5, Panel D)
Number analyzed (Participants) | 9 | 9 | 10 | 9 | 5
Participants
  Entire treatment period (48 Wks) | 3 | 4 | 4 | 1 | 1
  During TMC435/Placebo treatment (4 Wks) | 2 | 1 | 0 | 1 | 0
  During treatment with RBV and PegIFNα-2a (44 Wks) | 1 | 3 | 4 | 0 | 1

17. Secondary Outcome: Viral Relapse in Treatment-Naïve Hepatitis C Virus (HCV)-Infected Participants (Cohort 1 and 2, Panel A and B Combined)
Description: The table below shows the number of treatment-naïve participants with viral relapse (defined as having confirmed detectable plasma level of HCV ribonucleic acid [RNA] during the follow-up period in participants with undetectable plasma HCV RNA [less than 25 IU/mL undetectable] at the end of treatment) for the treatment groups in Cohort 1 (Panel A and B combined) and in Cohort 2 (Panel A and B combined). See "treatment-naïve" defined above.
Time Frame: Up to Week 72
Population: The analysis population used to evaluate viral relapse included participants in the intent-to-treat population (defined as all participants who were randomized and received at least one dose of study medication) who were treatment-naïve and had undetectable plasma HCV RNA (less than 25 IU/mL undetectable) at the end of treatment.
Measure: Number; unit: Participants
Groups:
- TMC435 75 mg (Cohort 1, Panel A and B): Treatment-naïve participants received TMC435 75 mg once daily for 7 days followed by TMC435 75 mg once daily coadministered with RBV for 21 days + PegIFNα-2a on Days 8, 15, and 22 (Panel A) OR TMC435 75 mg once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22 (Panel B).
- Placebo (Cohort 1, Panel A and B): Treatment-naïve participants received placebo (identical in appearance to TMC435 25 mg or 75 mg) once daily for 7 days followed by Placebo once daily coadministered with RBV for 21 days + peginterferon alpha-2a (PegIFNα-2a) on Days 8, 15, and 22 (Panel A) OR placebo once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22 (Panel B).
Arm/Group | TMC435 25 mg (Cohort 1, Panel A and B) | TMC435 75 mg (Cohort 1, Panel A and B) | Placebo (Cohort 1, Panel A and B) | TMC435 200 mg (Cohort 2, Panel A and B) | Placebo (Cohort 2, Panel A and B)
Number analyzed (Participants) | 15 | 18 | 12 | 14 | 5
Participants
  Relapse | 2 | 1 | 2 | 1 | 0
  No relapse | 12 | 17 | 10 | 13 | 5
  Missing follow-up | 1 | 0 | 0 | 0 | 0

18. Secondary Outcome: Viral Relapse in Treatment-Experienced Hepatitis C Virus (HCV)-Infected Participants (Cohort 4, Panel C and Cohort 5, Panel D)
Description: The table below shows the number of treatment-experienced participants combined (non-responders and relapsers, see defined above) with viral relapse, defined as having confirmed detectable plasma level of HCV ribonucleic acid (RNA) during the follow-up period in participants with undetectable plasma HCV RNA (less than 25 IU/mL undetectable) at the end of treatment who received TMC435 or placebo coadministered with ribavirin for 28 days + peginterferon alpha-2a (PegIFNα-2a) on Days 1, 8, 15, and 22.
Time Frame: Up to Week 72
Population: The analysis population used to evaluate viral relapse included participants in the intent-to-treat population (defined as all participants who were randomized and received at least one dose of study medication) who were treatment-experienced and had undetectable plasma HCV RNA (less than 25 IU/mL undetectable) at the end of treatment.
Measure: Number; unit: Participants
Groups:
- TMC435 200 mg (Cohort 5, Panel D): Treatment-experienced relapsers in Cohort 5, Panel D received TMC435 200 mg once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22.
Arm/Group | TMC435 75 mg (Cohort 4, Panel C) | TMC435 150 mg (Cohort 4, Panel C) | TMC435 200 mg (Cohort 4, Panel C) | Placebo (TMC435 75/150/200 mg) (Cohort 4, Panel C) | TMC435 200 mg (Cohort 5, Panel D)
Number analyzed (Participants) | 6 | 3 | 6 | 3 | 3
Participants
  Relapse | 3 | 0 | 1 | 3 | 0
  No relapse | 3 | 3 | 5 | 0 | 3

19. Secondary Outcome: Sustained Virologic Response (SVR) in Treatment-Naïve Hepatitis C Virus (HCV)-Infected Participants (Cohort 1 and 2, Panel A and B Combined)
Description: The table below shows the number of treatment-naïve participants with an SVR to treatment (defined as having an undetectable plasma level of HCV ribonucleic acid after the last planned dose of treatment) for the treatment groups in Cohort 1 (Panel A and B combined) and in Cohort 2 (Panel A and B combined). SVR was measured at 4, 8, 12, and 24 weeks after the last dose of treatment (SVR4, SVR8, SVR12, and SVR24, respectively). See "treatment-naïve" defined above.
Time Frame: SVR4 (Week 52), SVR8 (Week 56), SVR12 (Week 60), and SVR24 (Week 72)
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- TMC435 75mg (Cohort 1, Panel A and B): Treatment-naïve participants received TMC435 75 mg once daily for 7 days followed by TMC435 75 mg once daily coadministered with RBV for 21 days + PegIFNα-2a on Days 8, 15, and 22 (Panel A) OR TMC435 75 mg once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22 (Panel B).
- Placebo (Cohort 1, Panel A and B): Treatment-naïve participants received placebo (identical in appearance to TMC435 25 mg or 75 mg) once daily for 7 days followed by Placebo once daily coadministered with RBV for 21 days + PegIFNα-2a on Days 8, 15, and 22 (Panel A) OR placebo once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22 (Panel B).
Arm/Group | TMC435 25 mg (Cohort 1, Panel A and B) | TMC435 75mg (Cohort 1, Panel A and B) | Placebo (Cohort 1, Panel A and B) | TMC435 200mg (Cohort 2, Panel A and B) | Placebo (Cohort 2, Panel A and B)
Number analyzed (Participants) | 18 | 19 | 13 | 18 | 6
Participants
  SVR4 | 12 | 16 | 11 | 12 | 5
  SVR8 | 12 | 14 | 9 | 12 | 5
  SVR12 | 12 | 15 | 9 | 12 | 5
  SVR24 | 10 | 15 | 9 | 12 | 5

20. Secondary Outcome: Sustained Virologic Response (SVR) in Treatment-Experienced Hepatitis C Virus (HCV)-Infected Participants (Cohort 4, Panel C and Cohort 5, Panel D)
Description: The table below shows the number of treatment-experienced participants (non-responders and relapsers, see defined above) in each treatment group in Cohort 4, Panel C and in Cohort 5, Panel D with an SVR to treatment defined as having an undetectable plasma level of HCV ribonucleic acid after the last planned dose of the entire treatment regimen. SVR was measured at 4, 8, 12, and 24 weeks after the last dose of treatment (SVR4, SVR8, SVR12, and SVR24, respectively).
Time Frame: SVR4 (Week 52), SVR8 (Week 56), SVR12 (Week 60), and SVR24 (Week 72)
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- Placebo (TMC435 75/150/200 mg) (Cohort 4, Panel C): Treatment-experienced non-responders received Placebo once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22.
Arm/Group | TMC435 75 mg (Cohort 4, Panel C) | TMC435 150 mg (Cohort 4, Panel C) | TMC435 200 mg (Cohort 4, Panel C) | Placebo (TMC435 75/150/200 mg) (Cohort 4, Panel C) | TMC435 200 mg (Cohort 5, Panel D)
Number analyzed (Participants) | 9 | 9 | 10 | 9 | 5
Participants
  SVR4 | 2 | 3 | 4 | 1 | 3
  SVR8 | 1 | 3 | 4 | 0 | 3
  SVR12 | 1 | 3 | 5 | 0 | 3
  SVR24 | 1 | 3 | 5 | 0 | 3

21. Secondary Outcome: Maximum Plasma Concentration (Cmax) of TMC435 in Treatment-Naïve Hepatitis C Virus (HCV)-Infected Participants (Cohort 1 and 2, Panel A and B)
Description: The table below shows the mean (standard deviation) Cmax for treatment-naïve participants at selected time points who were treated with TMC435 for 7 days followed by TMC435 coadministered with ribavirin for 21 days + peginterferon alpha-2a (PegIFNα-2a) on Days 8, 15, and 22 (Panel A) and with TMC435 coadministered with ribavirin for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22 (Panel B). See "treatment-naïve" defined above. The number of participants analyzed at Day 28 in the 6 treatment groups listed below from left to right were 9, 8, 7, 9, 9, and 10.
Time Frame: Days 1 and 28 (predose and 0.5, 1, 2, 4, 6, 8, and 10 hours postdose)
Population: All participants who received treatment were included in the pharmacokinetic (PK) analysis, however, due to various reasons (ie, missing samples at certain time points, or exclusion of specific plasma concentrations from the PK analysis) not all PK parameters could always be calculated for each participant.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- TMC435 25 mg (Cohort 1, Panel B): Treatment-naïve participants received TMC435 25 mg once daily coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22.
Arm/Group | TMC435 25 mg (Cohort 1, Panel A) | TMC435 75 mg (Cohort 1, Panel A) | TMC435 200 mg (Cohort 2, Panel A) | TMC435 25 mg (Cohort 1, Panel B) | TMC435 75 mg (Cohort 1, Panel B) | TMC435 200 mg (Cohort 2, Panel B)
Number analyzed (Participants) | 9 | 10 | 8 | 9 | 8 | 10
ng/mL
  Day 1 | 251.1 (77.40) | 1008 (490.9) | 3369 (1760) | 239.6 (125.8) | 958.0 (448.9) | 3945 (2096)
  Day 28 | 307.1 (88.16) | 1058 (547.5) | 11180 (8522) | 329.4 (186.9) | 1609 (1310) | 10900 (6974)

22. Secondary Outcome: Maximum Plasma Concentration (Cmax) of TMC435 in Treatment-Experienced Hepatitis C Virus (HCV)-Infected Participants (Cohort 4, Panel C and Cohort 5, Panel D)
Description: The table below shows the mean (standard deviation) Cmax for treatment-experienced participants (non-responders and relapsers, see defined above) following treatment with TMC435 coadministered with ribavirin for 28 days + peginterferon alpha-2a (PegIFNα-2a) on Days 1, 8, 15, and 22. The number of participants analyzed at Day 28 in the 4 treatment groups listed below from left to right were 8, 8, 10, and 3.
Time Frame: Days 1 and 28 (predose and 0.5, 1, 2, 4, 6, 8, and 10 hours postdose)
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- TMC435 75 mg (Cohort 4, Panel C): Treatment-experienced non-responders received TMC435 75 mg once daily coadministered with ribavirin (RBV) for 28 days + peginterferon (PegIFNα-2a) on Days 1, 8, 15, and 22.
Arm/Group | TMC435 75 mg (Cohort 4, Panel C) | TMC435 150 mg (Cohort 4, Panel C) | TMC435 200 mg (Cohort 4, Panel C) | TMC435 200 mg (Cohort 5, Panel D)
Number analyzed (Participants) | 9 | 9 | 9 | 4
ng/mL
  Day 1 | 882.1 (273.2) | 2422 (919.0) | 2877 (1399) | 3870 (565.0)
  Day 28 | 1481 (879.6) | 4383 (2374) | 8452 (6112) | 12220 (2917)

23. Secondary Outcome: Predose Plasma Concentration (C0h) of TMC435 in Treatment-Naïve Hepatitis C Virus (HCV)-Infected Participants (Cohort 1 and 2, Panel A and B)
Description: The table below shows mean (standard deviation) of C0h of TMC435 at selected time points following treatment with TMC435 for 7 days followed by TMC435 coadministered with ribavirin for 21 days + peginterferon alpha-2a (PegIFNα-2a) on Days 8, 15, and 22 (Panel A) or with TMC435 coadministered with ribavirin for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22 (Panel B) in treatment-naïve participants (see "treatment-naïve" defined above).The number of participants analyzed at Day 28 in the 6 treatment groups listed below from left to right were 9, 9, 8, 9, 9, and 10.
Time Frame: Day 2 (predose) and Day 28 (predose and 0.5, 1, 2, 4, 6, 8, and 10 hours postdose)
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- TMC435 25 mg (Cohort 1, Panel B): Treatment-naïve participants received TMC435 25 mg coadministered with RBV for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22.
Arm/Group | TMC435 25 mg (Cohort 1, Panel A) | TMC435 75 mg (Cohort 1, Panel A) | TMC435 200 mg (Cohort 2, Panel A) | TMC435 25 mg (Cohort 1, Panel B) | TMC435 75 mg (Cohort 1, Panel B) | TMC435 200 mg (Cohort 2, Panel B)
Number analyzed (Participants) | 8 | 9 | 8 | 9 | 9 | 10
ng/ml
  Day 2 | 64.51 (37.57) | 209.3 (107.4) | 1053 (526.5) | 65.73 (41.75) | 281.6 (288.1) | 821.7 (422.9)
  Day 28 | 64.78 (35.15) | 331.6 (326.6) | 6913 (7726) | 95.83 (61.56) | 632.8 (1128) | 4818 (5071)

24. Secondary Outcome: Predose Plasma Concentration (C0h) of TMC435 in Treatment-Experienced Hepatitis C Virus (HCV)-Infected Participants (Cohort 4, Panel C and Cohort 5, Panel D)
Description: The table below shows mean (standard deviation) of C0h for treatment-experienced participants (non-responders and relapsers, see defined above) following treatment with TMC435 coadministered with ribavirin for 28 days + peginterferon alpha-2a (PegIFNα-2a) on Days 1, 8, 15, and 22. The number of participants analyzed at Day 2 and Day 28 differed as follows: At Day 2, the number of participants in the 4 treatment groups (from left to right) were 8, 7, 10, and 5; the number of participants analyzed at Day 28 in the 4 treatment groups (from left to right) were 9, 8, 10, and 4.
Time Frame: Day 2 (predose) and Day 28 (predose and 0.5, 1, 2, 4, 6, 8, and 10 hours postdose)
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TMC435 75 mg (Cohort 4, Panel C) | TMC435 150 mg (Cohort 4, Panel C) | TMC435 200 mg (Cohort 4, Panel C) | TMC435 200 mg (Cohort 5, Panel D)
Number analyzed (Participants) | 9 | 8 | 10 | 5
ng/mL
  Day 2 | 278.4 (192.2) | 733.6 (436.4) | 669.8 (301.7) | 1280 (955.8)
  Day 28 | 324.3 (351.9) | 1431 (1501) | 4145 (4425) | 5593 (3817)

25. Secondary Outcome: Average Steady-state Plasma Concentration (Css,av) of TMC435 in Treatment-Naïve Hepatitis C Virus (HCV)-Infected Participants (Cohort 1 and 2, Panel A and B)
Description: The table below shows mean (standard deviation)of Css,av for TMC435 in treatment-naïve HCV-infected participants at selected time points administered TMC435 for 7 days followed by TMC435 coadministered with ribavirin for 21 days + peginterferon alpha-2a (PegIFNα-2a) on Days 8, 15, and 22 (Panel A) and with TMC435 coadministered with ribavirin for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22 (Panel B). See "treatment-naïve" defined above. The number of participants analyzed at Day 28 in the 6 treatment groups listed below from left to right were 9, 8, 7, 9, 9, and 10.
Time Frame: Day 7 (predose); Day 28 (predose and 0.5, 1, 2, 4, 6, 8, and 10 hours postdose) (Panel A, Cohorts 1 and 2) and Day 28 (predose and 0.5, 1, 2, 4, 6, 8, and 10 hours postdose) (Panel B, Cohorts 1 and 2)
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- TTMC435 200 mg (Cohort 2, Panel A): Treatment-naïve participants received TMC435 200 mg once daily for 7 days followed by TMC435 200 mg once daily coadministered with RBV for 21 days + PegIFNα-2a on Days 8, 15, and 22.
Arm/Group | TMC435 25 mg (Cohort 1, Panel A) | TMC435 75 mg (Cohort 1, Panel A) | TTMC435 200 mg (Cohort 2, Panel A) | TMC435 25 mg (Cohort 1, Panel B) | TMC435 75 mg (Cohort 1, Panel B) | TMC435 200 mg (Cohort 2, Panel B)
Number analyzed (Participants) | 9 | 9 | 7 | 9 | 10 | 10
ng/ml
  Day 7 | 180.9 (90.04) | 832.3 (415.1) | 5714 (4157) | NA (NA) — Value not measured | NA (NA) — Value not measured | NA (NA) — Value not measured
  Day 28 | 170.4 (62.42) | 681.4 (414.7) | 7117 (6699) | 186.5 (115.7) | 986.0 (1087) | 7182 (5415)

26. Secondary Outcome: Average Steady-state Plasma Concentration (Css,av) of TMC435 in Treatment-Experienced Hepatitis C Virus (HCV)-Infected Participants (Cohort 4, Panel C and Cohort 5, Panel D)
Description: The table below shows mean (standard deviation) of Css,av for TMC435 in treatment-experienced HCV-infected participants (non-responders and relapsers, see defined above) at selected time points following treatment with TMC435 coadministered with ribavirin for 28 days + peginterferon alpha-2a (PegIFNα-2a) on Days 1, 8, 15, and 22.
Time Frame: Day 28 (predose and 0.5, 1, 2, 4, 6, 8, and 10 hours postdose)
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | TMC435 75 mg (Cohort 4, Panel C) | TMC435 150 mg (Cohort 4, Panel C) | TMC435 200 mg (Cohort 4, Panel C) | TMC435 200 mg (Cohort 5, Panel D)
Number analyzed (Participants) | 8 | 7 | 10 | 3
ng/ml | 820.8 (580.1) | 2435 (1909) | 6353 (5313) | 9613 (3981)

27. Secondary Outcome: Area Under the Plasma Concentration-time Curve From the Time of Administration to 24 Hours After Dosing (AUC24h) of TMC435 in Treatment-Naïve Hepatitis C Virus (HCV)-Infected Participants (Cohort 1 and 2, Panel A and B)
Description: The table below shows mean (standard deviation) values of the area under the plasma concentration-time curve from time of administration to 24 hours after dosing for TMC435 in treatment-naïve HCV-infected participants administered TMC435 for 7 days followed by TMC435 coadministered with ribavirin for 21 days + peginterferon alpha-2a (PegIFNα-2a) on Days 8, 15, and 22 (Panel A) and with TMC435 coadministered with ribavirin for 28 days + PegIFNα-2a on Days 1, 8, 15, and 22 (Panel B).The number of participants analyzed at Day 28 in the 6 treatment groups listed below from left to right were 9, 8, 7, 9, 9, and 10.
Time Frame: Days 1 and 28 (predose and 0.5, 1, 2, 4, 6, 8, and 10 hours postdose)
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | TMC435 25 mg (Cohort 1, Panel A) | TMC435 75 mg (Cohort 1, Panel A) | TMC435 200 mg (Cohort 2, Panel A) | TMC435 25 mg (Cohort 1, Panel B) | TMC435 75 mg (Cohort 1, Panel B) | TMC435 200 mg (Cohort 2, Panel B)
Number analyzed (Participants) | 9 | 10 | 8 | 9 | 8 | 10
ng.h/mL
  Day 1 | 3035 (1205) | 12240 (5663) | 43430 (22280) | 2853 (1207) | 12790 (7888) | 45700 (24160)
  Day 28 | 3961 (1523) | 16600 (10680) | 167200 (154500) | 4527 (2806) | 23610 (26780) | 169400 (126500)

28. Secondary Outcome: Area Under the Plasma Concentration-time Curve From the Time of Administration to 24 Hours After Dosing (AUC24h) of TMC435 in Treatment-Naïve Hepatitis C Virus (HCV)-Infected Participants (Cohort 4, Panel C and Cohort 5, Panel D)
Description: The table below shows mean (standard deviation) values of the area under the plasma concentration-time curve from time of administration to 24 hours after dosing for TMC435 in treatment-experienced HCV-infected participants considered non-responders (participants who achieved less than a 2 log10 IU/mL decline from baseline in plasma HCV ribonucleic acid (RNA) levels after 12 weeks of previous interferon [IFN]-based therapy [pegylated or non-pegylated]) or relapsers (defined as a participant with undetectable plasma HCV RNA at the end of treatment of previous IFN-based therapy and subsequent confirmed detectable plasma HCV RNA levels during follow-up at selected time points following treatment with TMC435 coadministered with ribavirin (RBV) for 28 days + peginterferon alpha-2a (PegIFNα-2a) on Days 1, 8, 15, and 22. The number of participants analyzed at Day 28 in the 4 treatment groups listed below from left to right was 8, 7, 10, and 3.
Time Frame: Days 1 and 28 (predose and 0.5, 1, 2, 4, 6, 8, and 10 hours postdose)
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | TMC435 75 mg (Cohort 4, Panel C) | TMC435 150 mg (Cohort 4, Panel C) | TMC435 200 mg (Cohort 4, Panel C) | TMC435 200 mg (Cohort 5, Panel D)
Number analyzed (Participants) | 9 | 9 | 9 | 4
ng.h/mL
  Day 1 | 11150 (2903) | 30920 (13450) | 34410 (14440) | 51300 (16720)
  Day 28 | 20150 (14720) | 57440 (44730) | 152600 (126600) | 231300 (96890)

ADVERSE EVENTS:
Time Frame: Up to 72 weeks.
Arm/Group | TMC435 25 mg (Cohort 1/Panel A and B) | TMC435 75mg (Cohort 1/Panel A and B) | Placebo (Cohort 1/Panel A and B) | TMC435 200 mg (Cohort 2, Panel A and B) | Placebo (Cohort 2/Panel A and B) | TMC435 75 mg (Cohort 4/Panel C) | TMC435 150 mg (Cohort 4/Panel C) | TMC435 200 mg (Cohort 4/Panel C) | Placebo (Cohort 4/Panel C) | TMC435 200 mg (Cohort 5/Panel D) | All TMC435 (All Cohorts)
Serious Adverse Events (participants affected / at risk) | 2/18 | 3/19 | 3/13 | 3/18 | 0/6 | 1/9 | 1/9 | 2/10 | 0/9 | 1/5 | 13/88
Other Adverse Events (participants affected / at risk) | 18/18 | 19/19 | 13/13 | 18/18 | 6/6 | 8/9 | 9/9 | 10/10 | 9/9 | 5/5 | 87/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TMC435 25 mg (Cohort 1/Panel A and B) (N=18) | TMC435 75mg (Cohort 1/Panel A and B) (N=19) | Placebo (Cohort 1/Panel A and B) (N=13) | TMC435 200 mg (Cohort 2, Panel A and B) (N=18) | Placebo (Cohort 2/Panel A and B) (N=6) | TMC435 75 mg (Cohort 4/Panel C) (N=9) | TMC435 150 mg (Cohort 4/Panel C) (N=9) | TMC435 200 mg (Cohort 4/Panel C) (N=10) | Placebo (Cohort 4/Panel C) (N=9) | TMC435 200 mg (Cohort 5/Panel D) (N=5) | All TMC435 (All Cohorts) (N=88)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Sinus arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cupulolithiasis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia escherichia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus insulin-dependent (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Toe deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Panic reaction (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Drug abuser (Social circumstances) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Social stay hospitalisation (Social circumstances) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TMC435 25 mg (Cohort 1/Panel A and B) (N=18) | TMC435 75mg (Cohort 1/Panel A and B) (N=19) | Placebo (Cohort 1/Panel A and B) (N=13) | TMC435 200 mg (Cohort 2, Panel A and B) (N=18) | Placebo (Cohort 2/Panel A and B) (N=6) | TMC435 75 mg (Cohort 4/Panel C) (N=9) | TMC435 150 mg (Cohort 4/Panel C) (N=9) | TMC435 200 mg (Cohort 4/Panel C) (N=10) | Placebo (Cohort 4/Panel C) (N=9) | TMC435 200 mg (Cohort 5/Panel D) (N=5) | All TMC435 (All Cohorts) (N=88)
Anaemia (Blood and lymphatic system disorders) | 3 | 2 | 3 | 5 | 1 | 3 | 1 | 2 | 0 | 0 | 16
Neutropenia (Blood and lymphatic system disorders) | 5 | 7 | 1 | 6 | 2 | 2 | 3 | 3 | 1 | 0 | 26
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 8
Vertigo (Ear and labyrinth disorders) | 4 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 7
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 7
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 7
Constipation (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 4 | 1 | 2 | 0 | 3 | 1 | 3 | 2 | 1 | 21
Dry mouth (Gastrointestinal disorders) | 3 | 4 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 9
Nausea (Gastrointestinal disorders) | 9 | 6 | 1 | 6 | 2 | 3 | 3 | 4 | 1 | 0 | 31
Toothache (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 3 | 2 | 1 | 2 | 2 | 1 | 0 | 1 | 0 | 1 | 10
Asthenia (General disorders) | 6 | 9 | 4 | 5 | 1 | 1 | 2 | 3 | 2 | 0 | 26
Chills (General disorders) | 2 | 2 | 3 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 6
Fatigue (General disorders) | 10 | 8 | 5 | 7 | 3 | 3 | 5 | 2 | 5 | 3 | 38
Influenza like illness (General disorders) | 6 | 5 | 2 | 4 | 2 | 3 | 1 | 5 | 1 | 4 | 28
Injection site erythema (General disorders) | 1 | 2 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 6
Injection site reaction (General disorders) | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 5
Irritability (General disorders) | 4 | 1 | 1 | 1 | 1 | 1 | 1 | 2 | 2 | 2 | 12
Pain (General disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 3
Performance status decreased (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pyrexia (General disorders) | 6 | 3 | 2 | 4 | 0 | 2 | 3 | 3 | 2 | 0 | 21
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 2 | 0 | 2 | 1 | 1 | 1 | 2 | 0 | 0 | 10
Body temperature increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 6 | 1 | 1 | 2 | 0 | 0 | 3 | 1 | 3 | 0 | 13
Decreased appetite (Metabolism and nutrition disorders) | 2 | 5 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 4 | 1 | 3 | 0 | 3 | 4 | 1 | 2 | 0 | 20
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 1 | 0 | 0 | 0 | 2 | 3 | 2 | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 4 | 4 | 4 | 1 | 1 | 0 | 1 | 3 | 1 | 15
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Disturbance in attention (Nervous system disorders) | 2 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 2 | 9
Dizziness (Nervous system disorders) | 3 | 1 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 4 | 10
Dysgeusia (Nervous system disorders) | 1 | 1 | 3 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 6
Headache (Nervous system disorders) | 13 | 11 | 6 | 3 | 4 | 5 | 7 | 3 | 6 | 4 | 46
Depression (Psychiatric disorders) | 6 | 3 | 0 | 4 | 1 | 0 | 0 | 1 | 1 | 0 | 14
Insomnia (Psychiatric disorders) | 3 | 2 | 3 | 4 | 1 | 0 | 2 | 1 | 3 | 0 | 12
Loss of libido (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Mood altered (Psychiatric disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Nervousness (Psychiatric disorders) | 3 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 4
Sleep disorder (Psychiatric disorders) | 4 | 1 | 1 | 2 | 0 | 0 | 2 | 1 | 1 | 0 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 7 | 4 | 1 | 3 | 2 | 3 | 1 | 3 | 0 | 19
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 3 | 1 | 1 | 2 | 2 | 4 | 0 | 0 | 18
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 3 | 6
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 6 | 2 | 2 | 0 | 2 | 3 | 1 | 1 | 0 | 17
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 9 | 2 | 3 | 1 | 0 | 2 | 0 | 2 | 1 | 20
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 2 | 2 | 1 | 2 | 0 | 7
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3 | 2 | 5 | 0 | 3 | 3 | 3 | 5 | 3 | 21
Pruritus generalised (Skin and subcutaneous tissue disorders) | 5 | 1 | 2 | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 10
Rash (Skin and subcutaneous tissue disorders) | 1 | 3 | 3 | 4 | 1 | 0 | 0 | 1 | 1 | 2 | 11
Urticaria localised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 4
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Sinus arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Inner ear inflammation (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abnormal sensation in eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Dry eye (Eye disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Eye oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Eye pain (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Photophobia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retinal vein occlusion (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Bowel sounds abnormal (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breath odour (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 4
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Gastric disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gingivitis (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Glossodynia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Intestinal functional disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lip haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Periodontitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sensitivity of teeth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Face oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Feeling cold (General disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Feeling hot (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site bruising (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Injection site injury (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Mucosal dryness (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Non-cardiac chest pain (General disorders) | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 4
Xerosis (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Abscess jaw (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 4
Candidiasis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 3
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Eyelid infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Furuncle (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Genital candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gingival abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Gingival infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral fungal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 4
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Periorbital infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 3
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 2
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 4
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Blood phosphorus decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood uric acid increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
ECG signs of myocardial ischaemia (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematocrit decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Heart rate irregular (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 4
Weight decreased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Joint ankylosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Muscle tightness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Amnesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intercostal neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Migraine with aura (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
Syncope (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Affective disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aggression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Alcoholism (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Dependence (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depressed mood (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 4
Depressive symptom (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Emotional disorder (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Impulsive behaviour (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Libido decreased (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Listless (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neurosis (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tearfulness (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epididymitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lichen planus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 3
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Phlebitis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Raynaud's phenomenon (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vasculitis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less